CLINICAL TRIAL: NCT03542214
Title: Calcium Electroporation for the Treatment of Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HGH-2017-026
Record Dates: First submitted 2018-01-29; First posted 2018-05-31 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer Stage IV
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Calcium electroporation treatment (Experimental): Experimental treatment with calcium electroporation for inoperabel colorectal cancer
  Interventions: Combination Product: Calcium electroporation

INTERVENTIONS:
Combination Product: Calcium electroporation — Patients with inoperable colorectal cancer will be treated with calcium electroporation

SUMMARY:
In this phase I study 6 patients with inoperable colorectal cancer is treated with calcium electroporation to establish safety and efficacy of the treatment.

DETAILED DESCRIPTION:
A total of 6 evaluable patients with inoperable colorectal cancer are expected to be included in the study and the time for inclusion of patients is estimated to be 1-2 years. All patients will have been offered the standard of care and all available alternatives before entering the protocol. Calcium electroporation will not be compared to other means of treatment.

All patients will be treated once, but in case of residual tumor tissue at follow-up, and if the investigator considers it safe, they will be offered re-treatment. A maximum of 3 treatments per patient will be conducted with an interval of minimum 4 weeks. The patients will be followed with regular examinations for 12 months, starting from first treatment day.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified colorectal tumor
* Conferred by multidisciplinary team (radiologists, surgeons and oncologists) discussing options possible for the patient, resulting in agreement that an endoscopic treatment with calcium electroporation should be offered to the patient.
* Treatment free interval of minimum 2 weeks.
* Thrombocytes ≥ 50 billions/l, INR >1,2. Medical correction is allowed, e.g. correction of elevated INR by means of vitamin K.
* Performance status ECOG/WHO ≤2
* Both men and women who are sexually active must use safe contraception (contraceptive coil, deposit injection of gestagen, subdermal implantation, hormonal vaginal ring or transdermal patch.)
* Trial subject ≥ 18 years.
* Trial subject must be able to understand the participants' information.
* Signed informed consent. The patients are considered participants in the study after signing of the informed consent.

Exclusion criteria:

* Coagulative disturbance that cannot be corrected
* Pregnancy or lactation (Pregnancy is ruled out in fertile women by an HCG test in a blood sample)
* Concurrent participation in other clinical trials that involve experimental drugs or participation in a clinical trial involving experimental drugs within 4 weeks prior to administration of the drug in this study.
* Treatment with bevacizumab within the last 4 weeks.
* Heavily inflamed colorectal mucus membrane with bleeding or ulcerations.
* Implanted colon stent
* Other clinical disease or previous treatments that make the investigator deem the patient unfit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Safety of the calcium electroporation procedure in colorectal cancer (registration of adverse events; CTCAE v4 will be used) | 12 months
  Safety will be assessed through registration of adverse events related to the treatment. Furthermore, CT scans and follow-up endoscopies are performed as a safety marker to exclude any perforations, bleeding or infections. CTCAE v4 will be used.

SECONDARY OUTCOMES:
Local response | 18 months
  Tumor biopsies will be analyzed regarding standard histology and immunologic infiltration (CD8/CD3 and PD-L1/PD1)
Systemic respons to calcium electroporation in colorectal cancer. | 12 months
  Blood samples will be collected. Multiplex cytokine analyses and transcriptional analyses will be performed. Furthermore cell adhesion assay will be performed. Additionally circulating tumor DNA will be measured as a marker for the tumor burden
Tumorregression | 12 months
  CT/MR scans are performed and analyzed according to RECIST-criteria

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, DMSc, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided